CLINICAL TRIAL: NCT02222415
Title: The Impact of Timed Protein Supplementation to Maximize the Skeletal Muscle Adaptive Response to Resistance Type Exercise Training in Healthy Young Men
Brief Title: Exercise Training in Healthy Young Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MEC 11-03-45
Record Dates: First submitted 2014-08-20; First posted 2014-08-21 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Gaining Skeletal Muscle Mass and Strength
Keywords: Muscle mass; Strength; Cross-sectional area; Protein
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Training + placebo drink (Placebo Comparator): Exercise + non-caloric placebo drink
  Interventions: Dietary Supplement: Exercise + Protein drink
- Exercise + Protein drink (Experimental): exercise + Drink containing Protein, Carbohydrates and Fat
  Interventions: Dietary Supplement: Exercise + Protein drink

INTERVENTIONS:
Dietary Supplement: Exercise + Protein drink

SUMMARY:
Resistance type exercise training has been shown to be a potent stimulus to increase skeletal muscle mass and strength in healthy men. Furthermore, timed protein intake is also known to affect the muscle adaptive response following exercise. Whether timed protein intake could augment the increase in muscle fiber size and/or satellite cell content following long-term exercise intervention remains to be established.

We hypothesize that protein supplementation before sleep, on both training and non-training days, during a 12 week resistance training program further increases type II muscle fibre cross sectional area when compared to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Healthy
* Age between 18 and 30 years
* BMI between 18.5 and 30 kg/m2
* Recreationally active, performing sports on a non-competitive basis between 2 and 5 hours p/wk
* Participants willing and able to give written informed consent and to understand, to participate and to comply with the biomedical research project requirements

Exclusion Criteria:

* HbA1C level above 6.5%
* Fasted blood glucose level above 7 mmol/L
* Serum creatinine level beneath 60 or above 120 µmol/L
* Participants with a recent history or current state of COPD
* Participants with a recent history or current state of rheumatoid arthritis
* Participants with a recent history or current state of musculoskeletal/orthopedic disorders
* Participants with a recent history or current state of renal disorder
* Participants with a recent history or current state of cognitive impairment
* Participants with orthopedic metal implants in the spine and/or upper/lower extremities
* Participants with lactose intolerance and/or dairy protein allergy
* Participants who are enrolled in an interventional biomedical research project or have received an investigational new drug or product with the last 30 days prior to screening.
* Participants on medication, including anticoagulants

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2011-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle fiber size | 12 weeks
  Skeletal muscle fiber size will be assessed by muscle biopsy sampling before, during and after the 12 wks intervention period.
  Muscle fiber size will be expressed in µm2

SECONDARY OUTCOMES:
Quadriceps cross-sectional area | 12 weeks
  Quadriceps cross-sectional area will be assessed by CT-scan before and after the 12 wks intervention period.
  Quadriceps cross-sectional area will be expressed in cm2
Whole body en regional body composition | 12 weeks
  Body composition (whole-body as well as regional) well be determined by DXA-scan performed before and after the 12 wks intervention period.
  Results will be expressed in kilograms
1RM strength | 12 weeks
  Maximum muscle strength will be assessed before, during and after 12 wks of exercise training by means of a 1 rep max test and will be expressed in kilograms.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Cermak NM, Res PT, de Groot LC, Saris WH, van Loon LJ. Protein supplementation augments the adaptive response of skeletal muscle to resistance-type exercise training: a meta-analysis. Am J Clin Nutr. 2012 Dec;96(6):1454-64. doi: 10.3945/ajcn.112.037556. Epub 2012 Nov 7. PMID 23134885
- [Background] Res PT, Groen B, Pennings B, Beelen M, Wallis GA, Gijsen AP, Senden JM, VAN Loon LJ. Protein ingestion before sleep improves postexercise overnight recovery. Med Sci Sports Exerc. 2012 Aug;44(8):1560-9. doi: 10.1249/MSS.0b013e31824cc363. PMID 22330017
- [Derived] Snijders T, Res PT, Smeets JS, van Vliet S, van Kranenburg J, Maase K, Kies AK, Verdijk LB, van Loon LJ. Protein Ingestion before Sleep Increases Muscle Mass and Strength Gains during Prolonged Resistance-Type Exercise Training in Healthy Young Men. J Nutr. 2015 Jun;145(6):1178-84. doi: 10.3945/jn.114.208371. Epub 2015 Apr 29. PMID 25926415